CLINICAL TRIAL: NCT03404401
Title: BLI4700-301: A Safety and Efficacy Comparison of BLI4700 Bowel Preparation Versus an FDA-approved Comparator in Adult Subjects Prior to Colonoscopy
Brief Title: A Safety and Efficacy Comparison of BLI4700 Bowel Prep Versus an FDA-approved Comparator in Adults Prior to Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI4700-301
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-05

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLI4700 Bowel Preparation (Experimental)
  Interventions: Drug: BLI4700
- FDA Approved Bowel Preparation (Active Comparator)
  Interventions: Drug: Polyethylene glycol bowel preparation

INTERVENTIONS:
Drug: BLI4700 — Oral bowel preparation
  Arms: BLI4700 Bowel Preparation
Drug: Polyethylene glycol bowel preparation — Oral bowel preparation
  Arms: FDA Approved Bowel Preparation

SUMMARY:
The objective of this study is to compare the safety and efficacy of BLI4700 bowel preparation to an FDA-approved bowel preparation as 2-day, split-dose bowel preparations prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
* 18 to 85 years of age (inclusive)
* If female, and of child-bearing potential, is using an acceptable form of birth control
* Negative serum pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastroparesis, gastric retention, bowel perforation, toxic colitis or megacolon.
* Subjects with ongoing severe, acute inflammatory bowel disease
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
* Subjects taking diuretics, anti-hypertensive medications, including angiotensin converting enzyme (ACE) inhibitors and Angiotensin II receptor blockers (ARBs), or chronic NSAIDs, that have not been stable for 30 days. NSAID use for occasional pain is not exclusionary.
* Subjects with uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 100 mmHg).
* Subjects taking antibiotics within 7 days of colonoscopy.
* Subjects with severe renal insufficiency (GFR < 30 mL/min/1.73m2).
* Subjects with known severe hepatic insufficiency (Child Pugh C)
* Subjects with cardiac insufficiency (NYHA Functional Classifications 3 or 4).
* Subjects with an abnormal and clinically significant physical examination or ECG finding at Visit 1.
* Subjects undergoing insulin therapy for any indication.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects undergoing colonoscopy for foreign body removal and/or decompression.
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects allergic to any preparation component.
* Subjects using drugs of abuse, including abused prescription medications.
* Subjects who are withdrawing from alcohol or benzodiazepines.
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (23):
- United States (23):
  - Braintree Research Site 212, Mobile, Alabama
  - Braintree Research Site 204, Tucson, Arizona
  - Braintree Research Site 209, Anaheim, California
  - Braintree Research Site 219, Chula Vista, California
  - Braintree Research Site 206, Los Angeles, California
  - Braintree Research Site 220, San Diego, California
  - Braintree Research Site 221, Inverness, Florida
  - Braintree Research Site 222, Jacksonville, Florida
  - Braintree Research Site 201, Palm Harbor, Florida
  - Braintree Research Site 224, Atlanta, Georgia
  - Braintree Research Site 215, Decatur, Georgia
  - Braintree Research Site 223, Lake Charles, Louisiana
  - Braintree Research Site 211, Monroe, Louisiana
  - Braintree Research Site 207, Hagerstown, Maryland
  - Braintree Research Site 218, Flowood, Mississippi
  - Braintree Research Site 210, Great Neck, New York
  - Braintree Research Site 214, Cincinnati, Ohio
  - Braintree Research Site 213, Portland, Oregon
  - Braintree Research Site 216, Columbia, South Carolina
  - Braintree Research Site 202, Franklin, Tennessee
  - Braintree Research Site 203, Jackson, Tennessee
  - Braintree Research Site 217, Ogden, Utah
  - Braintree Research Site 208, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Palma JA, Bhandari R, Cleveland MV, Mishkin DS, Tesoriero J, Hall S, McGowan J. A Safety and Efficacy Comparison of a New Sulfate-Based Tablet Bowel Preparation Versus a PEG and Ascorbate Comparator in Adult Subjects Undergoing Colonoscopy. Am J Gastroenterol. 2021 Feb 1;116(2):319-328. doi: 10.14309/ajg.0000000000001020. PMID 33165006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
Started (Safety population - all patients that took preparation.) | 281 | 271
Completed | 263 | 252
Not Completed | 18 | 19

BASELINE CHARACTERISTICS:
Population: safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation | Total
Number analyzed (Participants) | 281 | 271 | 552
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 193 | 183 | 376
  >=65 years | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.9) | 58.4 (11.6) | 57.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 152 | 310
  Male | 123 | 119 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 31 | 58
  Not Hispanic or Latino | 254 | 240 | 494
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 8 | 10 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 43 | 45 | 88
  White | 221 | 212 | 433
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7
Diabetic [Count of Participants; unit: Participants] — Subjects with medical history of diabetes
  Participants | 33 | 39 | 72
Renal Insufficiency (GFR < 60) [Count of Participants; unit: Participants] — Subjects with baseline GFR < 60 mL/min/1.73 m2
  Participants | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Successful Bowel Cleansing
Description: % of subjects with successful bowel preparation rated by colonoscopist on a 4 point scale (1=poor to 4=excellent)
Time Frame: Day of colonoscopy
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
Number analyzed (Participants) | 278 | 270
Participants | 257 | 241
Statistical Analysis 1: Comparison: BLI4700 Bowel Preparation vs FDA Approved Bowel Preparation; Test type: Non-Inferiority — Non-inferiority margin was set at 10%; p < 0.001, Cochran-Mantel-Haenszel

2. Other Pre Specified Outcome: Abdominal Distension (Solicited Reports)
Description: Percentage of patients who reported abdominal distension (with associated severity) when directly queried by study personnel, out of all patients that reported that event
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
Number analyzed (Participants) | 281 | 271
percentage of patients
  Mild | 68 | 71
  Moderate | 30 | 29
  Severe | 1 | 0

3. Other Pre Specified Outcome: Abdominal Pain (Solicited Reports)
Description: Percentage of patients who reported abdominal pain (with associated severity) when directly queried by study personnel, out of all patients that reported that event
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
Number analyzed (Participants) | 281 | 271
percentage of patients
  Mild | 65 | 71
  Moderate | 35 | 29
  Severe | 0 | 0

4. Other Pre Specified Outcome: Nausea (Solicited Reports)
Description: Percentage of patients who reported nausea (with associated severity) when directly queried by study personnel, out of all patients that reported that event
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
Number analyzed (Participants) | 281 | 271
percentage of patients
  Mild | 71 | 77
  Moderate | 27 | 23
  Severe | 2 | 0

5. Other Pre Specified Outcome: Vomiting (Solicited Reports)
Description: Percentage of patients who reported vomiting (with associated severity) when directly queried by study personnel, out of all patients that reported that event
Time Frame: 2 days
Measure: Number; unit: percentage of patients
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
Number analyzed (Participants) | 281 | 271
percentage of patients
  Mild | 48 | 46
  Moderate | 52 | 54
  Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | BLI4700 Bowel Preparation | FDA Approved Bowel Preparation
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/271
Serious Adverse Events (participants affected / at risk) | 0/281 | 2/271
Other Adverse Events (participants affected / at risk) | 1/281 | 4/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI4700 Bowel Preparation (N=281) | FDA Approved Bowel Preparation (N=271)
wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI4700 Bowel Preparation (N=281) | FDA Approved Bowel Preparation (N=271)
dizziness (Nervous system disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT03404401/Prot_SAP_000.pdf